CLINICAL TRIAL: NCT05798819
Title: A Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate GLS-010 Plus Platinum-containing Chemotherapy With or Without Bevacizumab as First-line Treatment for Persistent, Recurrent, or Metastatic Cervical Cancer
Brief Title: A Study of GLS-010 Plus Platinum-containing Chemotherapy±Bevacizumab as First-line Treatment for Persistent, Recurrent, or Metastatic Cervical Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guangzhou Gloria Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLS-010-32
Record Dates: First submitted 2022-12-26; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Persistent, Recurrent, or Metastatic Cervical Cancer
MeSH Terms: conditions — Recurrence | interventions — zimberelimab; Paclitaxel; Cisplatin; Carboplatin; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLS-010+chemotherapy± bevacizumab (Experimental): GLS-010 in combination with cisplatin or carboplatin and paclitaxel± bevacizumab
  Interventions: Drug: GLS-010; Drug: Placebo; Drug: paclitaxel; Drug: cisplatin; Drug: carboplatin
- Placebo+chemotherapy± bevacizumab (Placebo Comparator): Placebo in combination with cisplatin or carboplatin and paclitaxel± bevacizumab
  Interventions: Drug: Placebo; Drug: paclitaxel; Drug: cisplatin; Drug: carboplatin; Drug: bevacizumab

INTERVENTIONS:
Drug: GLS-010 — IV infusion
  Arms: GLS-010+chemotherapy± bevacizumab
Drug: Placebo — IV infusion
Drug: paclitaxel — IV infusion
Drug: cisplatin — IV infusion
Drug: carboplatin — IV infusion
Drug: bevacizumab — IV infusion
  Arms: Placebo+chemotherapy± bevacizumab

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase III study to evaluate GLS-010 plus platinum-containing chemotherapy with or without bevacizumab as first-line treatment for persistent, recurrent, or metastatic cervical cancer.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled phase III study，aimed to evaluate the efficacy and safety of GLS-010 plus platinum-containing chemotherapy with or without bevacizumab as first-line treatment for persistent, recurrent, or metastatic cervical cancer.All enrolled patients will be randomly divided into 2 groups and continuously treated until any event that meets the criteria for end of the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent form.
2. Women aged ≥ 18 and ≤ 75 years.
3. ECOG of 0 or 1.
4. Life expectancy ≥ 12 weeks.
5. Cervical cancer patients with histologically confirmed PD-L1 positive (CPS ≥ 1),.The histological types include squamous cell carcinoma, adenocarcinoma, or adenosquamous cell carcinoma.
6. No prior systemic therapy for persistent, recurrent or metastatic ([FIGO] Stage IVB) disease,not amenable to curative surgery or concurrent chemoradiotherapy.
7. At least one measurable tumor lesion per RECIST v1.1; lesions previously treated with radiotherapy or other loco-regional therapy are not considered as target lesions unless the lesion has unequivocal progression or the biopsy is obtained to confirm maligancy.
8. Subjects must have adequate organ function.
9. Female subjects of childbearing potential must have a negative serum pregnancy test prior to the first dose. Female subject of childbearing potential must use acceptable effective methods of contraception from screening and must agree to continue these precautions until 6 months after the last dose of study drug.

Exclusion Criteria:

1. Patients with the opportunity to be cured by surgery and radiotherapy.
2. Received with concurrent chemoradiotherapy, adjuvant chemotherapy,neo- adjuvant chemotherapy within 4 weeks prior to randomization.
3. Active central nervous system (CNS) metastasis.
4. Patients with other malignancies prior to randomization. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, transitional cell carcinoma of urothelial cancer, or carcinoma in situ (e.g. breast cancer) that have been cured are not excluded.
5. Has an active autoimmune disease that has required systemic treatment.
6. With active serious infections.
7. Subjects with HIV infection ,active hepatitis B virus infection, active hepatitis C virus infection,active tuberculosis infection,active syphilis .
8. Has not recovered adequately from toxicity and/or complications from surgery prior to randomization.
9. . .
10. Has a contraindication or hypersensitivity to any component of cisplatin, carboplatin, paclitaxel, or bevacizumab.
11. Have received any investigational treatment in other clinical trials within 4 weeks prior to randomization.
12. Pregnant or lactating women,or women may become pregnant during treatment.
13. Has had an allogeneic tissue/solid organ/ hematopoietic stem cells transplant.
14. History of nervous system and mental disease. History of drug abuse.
15. The patient is not suitable to participate the study in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | Up to 2 years
  OS is defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
progression-free survival (PFS) | Up to 2 years
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1.
Objective Response Rate (ORR) | Up to 2 years
  Proportion of subjects who have a complete or partial response relative to baseline based on RECIST 1.1 criteria.
Duration of Response (DOR) | Up to 2 years
  Measured from the date of partial or complete response to therapy until the cancer progresses based on RECIST v1.1 criteria.
Disease Control Rate (DCR) | Up to 2 years
  DCR defined as the proportion of subjects' response of CR, PR, or SD based on RECIST v1.1 criteria.
Time to Response（TTR） | Up to 2 years
  TTR defined as the time from the date of randomization to the date when the response criteria are first met, based on RECIST v1.1 criteria.
Number of subjects with adverse events (AEs) | From the time of signed informed consent to 90 days after end of treatment.
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment
Quality of life (QoL) | Up to 2 years
  EORTC QLQ-C30 will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No